CLINICAL TRIAL: NCT06254989
Title: Effectiveness of a Structured Aerobic Exercise Program in Cancer Survivors - A Pilot Study
Brief Title: Effectiveness of an Aerobic Exercise Program in Cancer Survivors.
Acronym: ESAP-CS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Holy Name Medical Center, Inc. (Other)
Responsible Party: Principal Investigator, George Miller, Chief of Surgical Oncology, Holy Name Medical Center, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-01-HN
Record Dates: First submitted 2024-01-29; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Aerobic Exercise
Keywords: Exercise; Cancer; Survivorship
MeSH Terms: conditions — Motor Activity; Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Aerobic Exercise — Participants will engage in aerobic exercise at HNH fitness at a minimum of 2 days a week for 12 weeks. Participants will have their daily step count collected via the Fitbit during this period. VO2 measurements will also be collected during active intervention using the UNCCRI protocol.
  The structured aerobic exercise program (Weeks 3-14) will entail 30 minutes of aerobic activity, 3 days a week, on the treadmill, at a goal of between 50 to 70% of predicted VO2 maximum heart rate. All structured aerobic program sessions will take place at Holy Name Health (HNH) Fitness and will be overseen by our collaborator and Director of Human Performance (Reg Grant). Exercise data will be recorded in the Technogym MyWellness cloud. Participants who drop out or discontinue attendance (defined as 4 consecutive sessions missed without notification of absence) before completion of the 12-week study intervention period will be replaced.

SUMMARY:
A prospective study of cancer survivor patients enrolling in a pilot aerobic exercise program. The total enrollment will be fifteen patients. The study timeline includes a screening period of 4 weeks, baseline period of 2 weeks, and active study intervention for 12 weeks. Study enrollment will continue until all 15 subjects are enrolled or up to 12 months, whichever comes first.

DETAILED DESCRIPTION:
Study Population: Adult cancer survivors within one year of completing cancer-directed therapy.

Study Objective: To determine the feasibility of a prescription exercise program in a cancer survivor population

Specific Objectives:

1. Quantify the number of patients who successfully enroll and complete the Program.
2. Determine a preliminary benefit, if any, of the program with regard to biometric parameters (change in systolic blood pressure, BMI, body composition, average step count, VO2 max), laboratory parameters (Hgb A1c, CRP, Lipid Profile, IL-6, Apolipoprotein B, Vitamin D-25-OH, Vitamin B12 and Folate), patient-reported wellness surveys (SEE, SRQ, Sleep Surveys).

Study Endpoints/Outcomes:

A. Percentage of participants who complete the Program. B. Change in systolic blood pressure C. Change in BMI D. Change in body composition E. Change in Average daily step count F. Change in predicted VO2 max F. Change in participant-reported wellness surveys (SEE, SRQ, and Sleep Surveys) G. Change in Circumference measurements (hip, waist, and neck) H. Improvement in laboratory parameters (Hgb A1c, CRP, Lipid profile, IL-6, Alipoprotein B, Vitamin D-25-OH, Vitamin B12, Folate) I. Cancer recurrence

Sample Size: Fifteen subjects

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 yr.) cancer survivor patients who completed treatment within the past year and are able to physically participate in the interventional aerobic exercise program.

Exclusion Criteria:

* Non-ambulatory individuals
* Inability to communicate in English
* Lack of transportation to/from appointments (Of note, language and transportation exclusion criteria are based on practical needs for this pilot study. If effective, services would be open to a broader array of patients).
* On medications (e.g., Ozempic, Tirzepatide) which induce prolonged weight loss.
* Patients who received cancer-directed therapy within the past month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-02-12 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of providing a structured in-person aerobic exercise intervention | 6 months
  To determine the feasibility of providing a structured in-person aerobic exercise training intervention to cancer survivor patients by determining the percentage of enrolled patients who complete the study.

SECONDARY OUTCOMES:
Weight in Lbs | 6 months
  Change in weight (Lbs) from baseline
Blood Pressure in mmHg | 6 months
  Change in blood pressure (mmHg) from baseline
Heart Rate in bpm | 6 months
  Change in Heart rate (bpm) from baseline
Body Mass Index (BMI) in Kg/m2 | 6 months
  Change in BMI from baseline. BMI will be calculated as weight (kg)/height (m2).
Predicted VO2 max in ml/kg/min | 6 months
  Change in predicted VO2 max from baseline calculated as the milliliters of Oxygen used per kg of body weight per minute
Percentage lean body mass | 6 months
  Change in lean body mass percentage from baseline
Percentage visceral fat | 6 months
  Change in visceral fat percentage from baseline
Percentage total body fat | 6 months
  Change in total body fat percentage from baseline
Hip circumference measurement in cm | 6 months
  Change in hip circumference measurements from baseline
Waist circumference measurement in cm | 6 months
  Change in waist circumference measurements from baseline
Neck circumference measurements in cm | 6 months
  Change in Neck circumference measurements from baseline
Laboratory Assessments of Nutrition, Glucose control and cardiovascular health | 6 months
  Change in laboratory Assessments of Nutrition, Glucose control and cardiovascular health
Average daily step count | 6 months
  Change in average daily step count from baseline

CONTACTS AND LOCATIONS:
Overall Officials: George Miller, MD, Principal Investigator — Holy Name Medical Center

IPD SHARING:
Plan to Share IPD: Undecided